CLINICAL TRIAL: NCT04877938
Title: ACTLIFE: is Active Life-style Enough for Health and Wellbeing in Elderly?
Brief Title: ACTLIFE: is Active Life-style Enough?
Acronym: ACTLIFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, prof. Federico Schena, Professor, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRIN 2017
Record Dates: First submitted 2020-11-16; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Sedentary Behavior
Keywords: Physical Activity; Echological Intevention; Older Adults
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: 1 group echological intervention
  1 group standard physical activity intervention
  1 control group
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will be awared of he group they belong. However, Invesitgators and Outcome assessors will not know the group each single participant belogns to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Echological Intervention (Experimental): A starting point for this 'Ecological-Exercise-Intervention'(EEI), would be to limit sitting time to no more than 2 hours/day, and to stand up and move after 30 minutes of continuous sitting. In accordance with several epidemiologic evidences light-intensity activities would be encouraged to substitute sedentary time (e.g., standing up while talking on the telephone, ironing while watching TV). Taking into consideration the guidance provided by ecologic models of health behavior evidences about specific constructs to guide EEI may be derived from behavioral research on physical activity.
  Interventions: Behavioral: Echolgical physical activity Intervention
- Standard Physical Activity Intervention (Active Comparator): People included in this group will be assigned to a standard physical activity program that will follow the guidelines of the American College of Sport and Medicine. The program will include moderate intensity aerobic and strength training, three times a week for a total amunt of 200 min of physical activity/week.
  Interventions: Behavioral: Echolgical physical activity Intervention
- Control group (No Intervention): Individuals included in this group will be asked to keep their life style,without taking part in any physical activity program.

INTERVENTIONS:
Behavioral: Echolgical physical activity Intervention — 'Ecological-Exercise-Intervention'(EEI), would be to limit sitting time to no more than 2 hours/day, and to stand up and move after 30 minutes of continuous sitting. In accordance with several epidemiologic evidences light-intensity activities would be encouraged to substitute sedentary time (e.g., standing up while talking on the telephone, ironing while watching TV).
  Arms: Echological Intervention; Standard Physical Activity Intervention

SUMMARY:
Sedentary lifestyles in modern obesogenic society produce several dysfunctions that cause chronic diseases in lederly population and this phenomenon is becoming a major public health problem. Regular physical activity has a profound effect on the expression of the potentials of human resilience, resulting in a decreased risk of chronic diseases. The identification of the biological mechanisms that are candidates for exercise-induced health benefits through biological pathways that are largely different from those targeted by common drugs, is highly relevant, since it might help to improve our knowledge of the pathophysiology of the chronic diseases in the sedentary population as well as to maximize the efficacy of physical activity interventions by implementing the best possible exercise dosage in older adults. For this purpose, the first aim of this project will be to identify the bioactive molecules and functional mechanisms that are candidates for exercise-induced health benefits. Moreover, in the view of more reliable, ecological and tailored approaches to counteract the problem of sedentary lifestyle, the second aim of this project will be to evaluate the effectiveness of an ecological exercise intervention in comparison to a traditional exercise intervention in sedentary elderly individuals.

DETAILED DESCRIPTION:
The first aim of this projects will be to identify the bioactive molecules and functional mechanisms that are candidates for exercise-induced health benefits through biological pathways that are largely different from those targeted by common drugs. In the view of more reliable, ecological and tailored approaches to counteract the pandemic problem of sedentary lifestyle in elderly population, the second aim of this project will be to evaluate the effectiveness of an ecological exercise intervention (EEI) in comparison to traditional exercise intervention (TEI) in sedentary older adults.

Introduction: Despite our society has developed several advances in technology and medicine, the human genetic framework is largely tailored to support the physical activity (PA) patterns of hunter-gatherer societies living 2.5 million years ago, for which food finding was obligatorily associated to PA. The energy expenditure of hunter-gatherers (1,500 kcal/day) is similar to 3h/day of moderate-to-vigorous PA (MVPA). Contrarily, technological improvements have influenced the dramatic drop in human PA levels: 1/3 of adults worldwide are currently inactive, and the endemic inactivity trend starts in early life. Indeed, sedentary behaviors in contemporary obesogenic environments trigger dysfunctions that cause chronic diseases and this phenomenon is becoming a major public health problem. Interestingly, regular PA has a profound effect on the expression of the potentials of human resilience, resulting in numerous positive adaptations and decreased risk of chronic diseases.

Protective role of exercise on cardiovascular disease risk factors: There is strong epidemiological evidence indicating that regular PA is associated with reduced rates of cardiovascular disease (CVD), hypertension, stroke, metabolic syndrome and Type 2 diabetes. Moreover, a dose-response of PA is usually observed in the general population. It is important to note, that exercise training has an improving effect on endothelial function.

The polypill-like effect of Exercise: Despite, in the last 40 years the pandemic increase of cardio-metabolic diseases has paralleled the advances in medicine, CVD remains the leading cause of death worldwide. In this complicated scenario, Wald and Law first described a combination pill for CVD prevention, which they called a "polypill". These authors claimed that CVD could be reduced by 88% and strokes by 80% if all those over 55 years of age were given a polypill containing statin, low-dose aspirin, and folic acid. This controversial and provocative approach of "medicalizing" the population is not possible and not ethical, but polypill-like benefits are achievable with a drug-free intervention, regular PA. It is worth of mention that the identification of the bioactive molecules and biological mechanisms that are candidates for exercise-induced health benefits through biological pathways that are largely different from those targeted by common drugs, is highly relevant, since it might help to improve our knowledge of the pathophysiology of the chronic diseases in the sedentary eldely population as well as to maximize the efficacy of PA interventions by implementing the best possible exercise dosage, resulting in optimal circulating levels of "health" molecules.

The exercise polypill: Skeletal-muscle fibers can produce a plethora of secreted factors, including proteins, growth factors, cytokines, with such secretory capacity increasing during active exercise, myogenesis and muscle remodeling. Muscle-derived molecules exerting either paracrine or endocrine effects are termed "myokines" and can be consider the exercise polypill.

Since regular exercise has protective effects on cardiovascular diseases and, interestingly, it is more protective than expected based on the improvement of traditional risk factors (blood lipids, hypertension, diabetes) it is easy to speculate that additional positive effects could be mediated by myokines on targets such as adipose tissue or liver.

For example, IL-6 is probably the myokine prototype because its level increases with exercise intensity and duration. Systemic low-level inflammation is a cardinal feature of cardio-metabolic diseases, and it can be attenuated by the cumulative effect of regular exercise bouts, during which the muscle releases IL-6 which creates a healthy milieu by inducing the production of other anti-inflammatory cytokines. Another prototype of contraction-induced myokine is IL-15, with resistance exercise stimulating its secretion. Muscle-derived IL-15 is one of the mediators of the anti-obesity effects of exercise. Recent research identified a novel PGC-1 -induced myokine called iriscin. Iriscin is associated with improved aerobic fitness in cardiac patients, muscle mass, and metabolic factors in healthy people, and neurogenesis in animal models. Secreted protein acidic and rich in cysteine (SPARC) is a matricellular glycoprotein released into the bloodstream by skeletal muscle in response to aerobic exercise plays a pivotal role in adipocyte differentiation and adipose tissue turnover.

Myostatin, is a potent muscle-growth inhibitor, endurance or resistance exercise downgrade myostatin expression.

Another class of molecules which are potentially up-regulated with regular exercise and could have additional effects on the protective effects of regular exercise are neurotrophins. Among them, brain-derived neurotrophic factor (BDNF) is the most affected by exercise. Increased levels of BDNF are well documented, providing mechanistic support for a beneficial exercise effect in cognitive function. Furthermore, BDNF increases phosphorylation enhancing fatty acid oxidation and glucose utilization in skeletal muscle.The emerging general feature is that During physical inactivity, adipose tissue secretes pro-inflammatory cytokines, which can lead to development of metabolic and cardiovascular diseases, such as T2DM and atherosclerosis (Iyer et al., 2010). The study of myokines as potential biomarkers for effectiveness of exercise is an attractive approach to develop better physical protocols to apply to the elderly population.

Intervention approaches: Sedentary behaviors in older adults are strongly associated with systemic dysfunctions that cause chronic diseases and this phenomenon is becoming a major public health problem. Moreover, the recognized polypill-like effect of exercise, needs further research in order to identify the biological mechanisms that are candidates for exercise-induced health benefits. Furthermore, it is necessary to maximize the efficacy of PA interventions by implementing the best possible exercise dosage. In this complicated scenario, Owen and colleagues explain in their scientific contribution "Adults' Sedentary Behavior Determinants and Interventions" the relevant phases of the behavioral epidemiology research strategy on sedentary behavior for children and adults, highlighting several strengths of the evidence relevant to interventions and public health initiatives.

Ecological-Exercise-Intervention: One of the goals of public health interventions would be to reduce total sedentary time and also to increase the number of breaks in sedentary time. A starting point for this 'Ecological-Exercise-Intervention'(EEI), would be to limit sitting time to no more than 2 hours/day, and to stand up and move after 30 minutes of continuous sitting. In accordance with several epidemiologic evidences light-intensity activities would be encouraged to substitute sedentary time (e.g., standing up while talking on the telephone, ironing while watching TV). Taking into consideration the guidance provided by ecologic models of health behavior evidences about specific constructs to guide EEI may be derived from behavioral research on physical activity. However, further studies are needed to clarify the feasibility, acceptability, and effectiveness of EEI in young and adult populations. On this matter, promising results have been observed in studies targeting increases in daily walking. Moreover, systematic evaluations of these "natural approaches" could be highly informative, especially through assessing whether changes in sedentary time actually do result.

ELIGIBILITY:
Inclusion Criteria:

* for sedentary individuals: ≤700 METs/week measured by IPAQ
* for active individuals: ≥1000 METs/week measured by IPAQ

Exclusion Criteria:

* Presence of cardiovascular and respiratory diseases
* Presence of Hypertension
* Presence of neurodegenerative diseases
* Pesence of acuteor chronic conditions that might influence inlfammatory response
* Any vascular Diabetes-related complication
* Drugs or alchol abuse
* Presence of other health-related condition that might affect the practice of physical activity.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-06-20 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Measure of strandars healthy-related biochemical parameters | through study completion, an average of 8 months
  Blood samples will be collected two times: 1) between 7:00 and 9:00 am, following overnight fasting, 48h distant from the last exercise session and 2) immediately after a training session. After centrifugation, they will be divided in different aliquots of appropriate amount and stored a -80°C in order to: measure triglycerides, total cholesterol, blood glucose, aspartate transaminase, alanine transaminase, creatinine

SECONDARY OUTCOMES:
Measure of Daily Energy Expenditure | through study completion, an average of 8 months
  Each participant will be outfitted with an Actiheart device allowing heart rate and acceleration data to be simultaneously recorded 24 hours a day for 7 consecutive days.
  Health-related quality of life: The Italian version of the SF-36 health survey will be administrated before and after the interventions.
Measure of the appendicular muscle mass | through study completion, an average of 8 months
  Magnetic resonance imaging (MRI) will be performed using a 1.5 Tesla MRI system. T1-weighted images of the lower limbs will be acquired supine with the legs extended. On the basis of a signal-intensity threshold, muscle borders will be selected to delineate and differentiate muscle, fat, and connective tissue. In the thighs area, the vastus lateralis (VL), vastus medialis, vastus intermedius, and rectus femoris will be traced in each image and in combination made up the quadriceps. Quadriceps muscle volumes will be calculated by summing the areas of all the slices.
Measure of Musle architecture | through study completion, an average of 8 months
  In the thigh, sagittal ultrasound images of the VL muscle will be recorded with a GE ultrasound system (GE Logiq-7) equipped with an 8-12 MHz linear transducer. Images will be obtained with a 90° flexion of hip and knee, at 50% of femur length corresponding to the mid-belly of the VL muscle. The pennation angle of the VL fascicles will be measured as the angle between the VL muscle fascicles and the deep aponeurosis of the insertion.
Measure of systemic vascular function | through study completion, an average of 8 months
  The passive limb movement protocol consisted of 60 s of resting baseline femoral blood flow data collection, followed by 60 s of passive knee extension and flexion with the same measure. Blood velocity will be analyzed with 1 Hz resolution on the Doppler ultrasound system (GE Logiq-7) for 60 s at rest and second by second for the first 60 s following the initiation of PLM.
Measure of cirulating level of hormones | through study completion, an average of 8 months
  Blood samples will be collected two times: 1) between 7:00 and 9:00 am, following overnight fasting, 48h distant from the last exercise session and 2) immediately after a training session. After centrifugation, they will be divided in different aliquots of appropriate amount and stored a -80°C in order to: measure cirulatin glevels of hormones such as: GH, IGF-1, IGFBP3, insulin and cortisol; the pro- and anti-inflammatory markers, C Reactive Protein (CRP), IL-1, IL-6 and IL-1ra; and of the sex-hormones testosterone, oestradiol, oestrone and sex hormone-binding globulin (SHBG);
Measure of cirulating bioactive markers | through study completion, an average of 8 months
  Blood samples will be collected two times: 1) between 7:00 and 9:00 am, following overnight fasting, 48h distant from the last exercise session and 2) immediately after a training session. After centrifugation, they will be divided in different aliquots of appropriate amount and stored a -80°C in order to measure circulating miRNA, PGC-1, Myonectin, Musclin, Sparc, Myostatin, BDNF, VEGF, and BDNF
Measure of cardio-metabolid health | through study completion, an average of 8 months
  Measurements of blood pressure will be performed with standard auscultatory and mercury sphygmomanometer technique.
  From a fasted venous blood sample Glucose, high- and low-density lipoprotein will be measured on a Cobas c501 (Roche Diagnostics GmbH, Mannheim, Germany), using proprietary reagents.
  Body anthropometrics will be measured with a standard protocol: body mass, height, body mass index calculation (BMI = body mass / height2), percent of body fat (7 skinfolds approach), waist and hip circumferences.
Measure of exercise capacity | through study completion, an average of 8 months
  To determine exercise capacity the subjects will perform an incremental walking maximal exercise trial (rest, 25%, 50%, 75%, and 100% of maximal exercise capacity). Breath-by-breath O2 expiratory airflow will be continuously recorded at rest, and during the exercise trial.
Measure of Lower limbs neuromuscular control | through study completion, an average of 8 months
  The force and EMG envelope rate of development during a maximum voluntary contraction and a tetanic stimulation will be compared in order to estimate the role of central command flow to the muscle in changing the efficiency of the tension development at the tendon. The maximal voluntary contraction will be started after a visual command will be done.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fiuza-Luces C, Garatachea N, Berger NA & Lucia A. (2013). Exercise is the real polypill. Physiology (Bethesda) 28, 330-358. Gilson ND, Ainsworth B, Biddle S, Faulkner G, Murphy MH, Niven A, Pringle A, Puig-Ribera A, Stathi A & Umstattd MR. (2009a). A multi-site comparison of environmental characteristics to support workplace walking. Prev Med 49, 21-23. Gilson ND, Puig-Ribera A, McKenna J, Brown WJ, Burton NW & Cooke CB. (2009b). Do walking strategies to increase physical activity reduce reported sitting in workplaces: a randomized control trial. Int J Behav Nutr Phys Act 6, 43. Iyer A, Fairlie DP, Prins JB, Hammock BD & Brown L. (2010). Inflammatory lipid mediators in adipocyte function and obesity. Nat Rev Endocrinol 6, 71-82. Joyner MJ & Green DJ. (2009). Exercise protects the cardiovascular system: effects beyond traditional risk factors. J Physiol 587, 5551-5558. Knaepen K, Goekint M, Heyman EM & Meeusen R. (2010). Neuroplasticity - exercise-induced response of peripheral brain-derived neurotrophic factor: a systematic review of experimental studies in human subjects. Sports Med 40, 765-801. Louis E, Raue U, Yang Y, Jemiolo B & Trappe S. (2007). Time course of proteolytic, cytokine, and myostatin gene expression after acute exercise in human skeletal muscle. J Appl Physiol (1985) 103, 1744-1751. Matthews CE, George SM, Moore SC, Bowles HR, Blair A, Park Y, Troiano RP, Hollenbeck A & Schatzkin A. (2012). Amount of time spent in sedentary behaviors and cause-specific mortality in US adults. Am J Clin Nutr 95, 437-445. Owen N, Sugiyama T, Eakin EE, Gardiner PA, Tremblay MS & Sallis JF. (2011). Adults' sedentary behavior determinants and interventions. Am J Prev Med 41, 189-196. Riechman SE, Balasekaran G, Roth SM & Ferrell RE. (2004). Association of interleukin-15 protein and interleukin-15 receptor genetic variation with resistance exercise training responses. J Appl Physiol (1985) 97, 2214-2219. Sallis JF, Cervero RB, Ascher W, Henderson KA, Kraft MK & Kerr J. (2006). An ecological approach to creating active living communities. Annu Rev Public Health 27, 297-322. Venturelli M, Pedrinolla A, Boscolo Galazzo I, Fonte C, Smania N, Tamburin S, Muti E, Crispoltoni L, Stabile A, Pistilli A, Rende M, Pizzini FB & Schena F. (2018). Impact of Nitric Oxide Bioavailability on the Progressive Cerebral and Peripheral Circulatory Impairments During Aging and Alzheimer's Disease. Frontiers in Physiology 9. Wald NJ & Law MR. (2003). A strategy to reduce cardiovascular disease by more than 80%. BMJ 326, 1419. Walther C, Gaede L, Adams V, Gelbrich G, Leichtle A, Erbs S, Sonnabend M, Fikenzer K, Korner A, Kiess W, Bruegel M, Thiery J & Schuler G. (2009). Effect of increased exercise in school children on physical fitness and endothelial progenitor cells: a prospective randomized trial. Circulation 120, 2251-2259.